CLINICAL TRIAL: NCT03381365
Title: A Pilot Study to Assess the Efficacy of an Anorectal Fistula Plug With Sealing of the Internal Opening (Curaseal AF) as a Treatment for Perianal Fistula
Brief Title: Efficacy of an Anorectal Fistula Plug With Sealing of the Internal Opening as a Treatment for Perianal Fistula
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 195923
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2017-09

CONDITIONS: Fistula in Ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- investigational arm (Experimental)
  Interventions: Device: CuraSeal Percutaneous Intraluminal Closure System

INTERVENTIONS:
Device: CuraSeal Percutaneous Intraluminal Closure System

SUMMARY:
The investigators aim to assess the efficacy of the Curaseal anal plug in patients with idiopathic uncomplicated fistulous tracts. Healing of the fistula tract will be assessed both clinically and radiologically with MR imaging.

DETAILED DESCRIPTION:
Perianal fistula is a challenging condition for colorectal surgeons. Achieving a favourable balance between healing and incontinence is the key to success. Surgeons have adopted many methods to close off this abnormal tract, which include laying opening, use of setons, advancement flaps and permanent stoma. A more recent approach has been the use of devices or substances to block the tract in the hope that it will seal off. Most of the devices that have been used to close the tract have not proved to be as effective in healing as a lay open with high rates of fistula persistence. A major failure of the devices has been their early expulsion and their inability to seal off the internal opening.

The new Curaseal plug may be able to overcome these shortcomings. This plug has a disc to seal the internal opening, with a suture to be placed at the external opening, which may prevent it falling out and ensure internal opening closure.

The investigators aim to assess the efficacy of the Curaseal anal plug in patients with idiopathic uncomplicated fistulous tracts. Healing of the fistula tract will be assessed both clinically and radiologically with MR imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are psychologically stable and suitable for intervention and able to provide informed consent

  * Patients who are willing and competent to fill in questionnaires and undergo investigations at various time points during the study
  * Patients with an idiopathic extra and trans-sphincteric perianal fistula.

Exclusion Criteria:

* Patients aged less than 18 or >80 years.
* Patients unfit to undergo general or spinal anaesthesia.
* Patients with a supra-levator fistula.
* Patients with a rectovaginal fistula.
* Patients with inflammatory bowel disease (Crohn's disease, ulcerative colitis).
* Patients with a fistula secondary to trauma, foreign body, developmental cyst or pelvic irradiation.
* Patients who are immunosuppressed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
fistula healing | 1 year
  clinical and radiological healing

SECONDARY OUTCOMES:
adverse effects or perioperative compilations related to device | within first year

CONTACTS AND LOCATIONS:
Locations (1):
- London North West Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No